CLINICAL TRIAL: NCT01891916
Title: Preventive Effect of Lactobacillus GG on Atopic Manifestation in Children With Cow's Milk Allergy
Brief Title: Effect Of Lactobacillus GG on Atopic March
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109/11
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Cow's Milk Allergy; Atopic Disease
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- extensively hydrolysed casein formula (No Intervention): extensively hydrolysed casein formula
- Extensively hydrolyzed casein formula + LGG (Active Comparator): Extensively hydrolized formula plus LGG
  Interventions: Dietary Supplement: Extensively hydrolyzed casein formula + LGG

INTERVENTIONS:
Dietary Supplement: Extensively hydrolyzed casein formula + LGG — Extensively hydrolyzed formula containing Lactobacillus GG
  Other Names: Extensively hydrolyzed formula plus LGG
  Arms: Extensively hydrolyzed casein formula + LGG

SUMMARY:
Food allergy (FA), defined as an adverse immune response to food allergens, is among the most frequent allergic disorders in childhood and it has recognized as a major paediatric health problem due to the severity of the reactions and the dramatic increase over the past decades. Cow's milk allergy (CMA) is the most frequent FA in children worldwide, and it has been demonstrated that it could be the first manifestation of the so-called "atopic march", characterized by the occurrence of other allergic disorders in the subsequent years after the onset of CMA. In a previous study, involving children with CMA over a period of 5 years, 40% developed asthma, 21% atopic eczema, and 43% allergic rhinitis. Similar results have been reported in a recent study on Finnish children Intestinal microflora appears to have a crucial role in the development of atopic disorders. Children with atopic diseases have different commensal bacterial groups in the gut compared to non-atopic children, and differences are also found between countries with high and low incidence of atopic diseases. There is currently great interest in manipulating the normal microbiota to accrue health benefits through an approach known as "probiotics." Probiotics are defined as "live microorganisms which when administered in adequate amounts confer a health benefit on the host". The conceptual basis of possible use of probiotics in the prevention and treatment of atopic disorders is well grounded. Lactobacillus GG (LGG) is the most studied probiotic in the prevention and treatment of atopic disorders. Wide and well-designed clinical studies have provided several evidences on the efficacy of LGG as preventive or therapeutic strategy in pediatric atopic disorders. More recently, in vitro studies have provided evidences on the potent immunoregulatory role and on the influence on intestinal microflora composition (toward a more beneficial composition in the prevention and treatment of atopic disorders) elicited by LGG. This view has been further reinforced by recent research showing that LGG is able to improve recovery of intestinal symptoms in infants with CMA-induced allergic colitis.

ELIGIBILITY:
Inclusion Criteria:

* infants aged less than 12 months, with a diagnosis of cow's milk allergy

Exclusion Criteria:

* age higher than 12 months,
* concomitant chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal tract,
* suspected eosinophilic esophagitis or eosinophilic enterocolitis,
* suspected food-protein-induced enterocolitis syndrome,
* suspected cow's milk proteins-induced anaphylaxis

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2008-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of allergic manifestations | 3 yrs
  Occurrence of allergic manifestations in children with CMA including atopic eczema, allergic urticaria, asthma, allergic rhinitis.Information on social and demographic factors, family and living conditions, and smoking habits will be documented. Unscheduled visit will be made when possible allergic symptoms will appear. Every 12 months sensitization to common dietary and respiratory antigens will be assessed by skin prick tests (SPT) and prick by prick tests.

SECONDARY OUTCOMES:
Allergic sensitization | 3 yrs
  Every 12 months sensitization to common dietary and respiratory antigens will be assessed by skin prick tests (SPT) and prick by prick tests.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy